CLINICAL TRIAL: NCT06923839
Title: Testing the Potential Metabolic Effect of the Human Gut Bacterial Peptide, RUCILP, in Healthy Men
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oluf Pedersen (Other)
Responsible Party: Sponsor-Investigator, Oluf Pedersen, Professor, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-22011935
Record Dates: First submitted 2025-03-20; First posted 2025-04-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-04

CONDITIONS: Healthy Male Adults
Keywords: Metabolism; Duodenal infusion; Postbiotics; Gut bacterial peptide; Intervention study; Intestinal infusion; Ruminococcus torques; Plasma glucose; Plasma insulin; Plasma PYY; Plasma incretins; Plasma GIP; Plasma RUCILP; Plasma GLP-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparator that is identical to the active arm except for the absence of RUCILP
  Interventions: Other: Placebo
- Active (Active Comparator): Intervention is identical to the placebo arm except for the addition of RUCILP to the infusion.
  Interventions: Biological: Test bacterial peptide: RUCILP

INTERVENTIONS:
Biological: Test bacterial peptide: RUCILP — The naturally occuring gut peptide RUCILP synthesized by the commensal gut bacterium Ruminococcus torques
  Arms: Active
Other: Placebo — Placebo is identical to the active intervention except for the absence of the RUCILP molecule.
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blinded and placebo-controlled clinical cross-over trial is in healthy men to explore the potential metabolic effects of the naturally occurring gut bacterial polypeptide, RUCILP. This bacterial peptide is produced by commensal strains of Ruminococcus torques in the human gut microbiota.

In preclinical studies of rodents, RUCILP lowers blood glucose and stimulates release of plasma insulin, glucagon-like peptide-1(GLP-1) and Peptide YY (PYY) but induces a decline of glucose-dependent insulinotropic polypeptide (GIP).

In the present trial, the investigators want to explore potential effects of intraduodenally delivered RUCILP on release of plasma concentrations of GLP-1, GIP and PYY.

In addition, the investigators will test for potential effects of intestinal RUCILP infusion on plasma concentrations of glucose, insulin and metabolome.

Participants will have a duodenal tube placed into which RUCILP or placebo will be infused over 3 hours after an initial standardized liquid meal infusion into the duodenal tube.

Participants will on different days and in a randomized order receive either placebo or RUCILP infusion into the tube.

Safety is acutely monitored under the intervention and postintervention safety is monitored by clinical biochemistry measures of hematology, and liver and kidney functions. The study participants will further keep a diary of any experienced adverse effects during the week after the intervention.

Primary OUTCOMES: a composite of changes in plasma concentrations of GLP-1, GIP and PYY.

Secondary OUTCOMES: changes in plasma glucose, plasma insulin and plasma metabolome profile.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Self-reported good health
* Caucasian
* Normal body mass index (18.5 to <25)

Exclusion Criteria:

* Any known disorder/disease that could interfere with study results or is seen as compromising to the study (as assessed by the investigator), for example diabetes, cancer or cardiovascular or kidney disease.
* Use of any daily medication as well as p.r.n. (pro re nata; not taken regularly) medication that cannot be discontinued during the trial
* Use of antibiotics during the recent three months
* Acute or chronic gastrointestinal symptoms
* Lactose intolerance
* Smoking
* Alcohol or drug abuse
* Use of creatine as dietary supplement during study period
* Plasma creatinine concentration above the normal range (>105 μmol/L)
* Known significant liver disease or plasma ALAT concentration ≥ 3 × normal value
* Values for hemoglobin, leukocytes, or thrombocytes outside of the normal ranges

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of GIP | During the 3 hours of RUCILP/placebo infusion
  Plasma measurements of GIP at different time points during the study day.
Plasma concentrations of GLP-1 | During the 3 hours of RUCILP/placebo infusion
  Plasma measurements of GLP-1 at different time points during the study day.
Plasma concentrations of PYY | During the 3 hours of RUCILP/placebo infusion
  Plasma measurements of PYY at different time points during the study day.

SECONDARY OUTCOMES:
Plasma concentrations of insulin | During the 3 hours of RUCILP/placebo infusion
  Plasma measurements of insulin at different time points during the study day.
Plasma concentrations of glucose | During the 3 hours of RUCILP/placebo infusion
  Plasma measurements of glucose at different time points during the study day.
Plasma metabolome profile | During the 3 hours of RUCILP/placebo infusion
  Plasma metabolome profile at different time points during the study day.
Plasma concentrations of RUCILP | During the 3 hours of RUCILP/placebo infusion
  Plasma measurements of RUCILP at different time points during the study day.

OTHER OUTCOMES:
Blood leukocytes | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of leukocytes in blood
Blood eosinophils | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of eosinophils in blood
Total blood leukocytes | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of total leukocytes in blood
Blood neutrophils | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of neutrophils in blood
Blood platelets | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of platelets in blood
Blood hemoglobin | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of hemoglobin in blood
Plasma alanine transaminase (ALT) | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of alanine transaminase (ALT) in plasma
Plasma aspartate transferase (AST) | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of aspartate transferase (AST) in plasma
Plasma alkaline phosphatase | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of alkaline phosphatase in plasma
Plasma albumin | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of albumin in plasma
Plasma creatinine | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of creatinine in plasma
Estimated Glomerular Filtration Rate (eGFR) | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
Plasma sodium | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of sodium in plasma
Plasma potassium | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of potassium in plasma
Plasma calcium (total) | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of total calcium in plasma
Plasma phosphate | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of phosphate in plasma
Plasma creatine kinase | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of creatine kinase in plasma
Plasma C-reactive protein | At baseline, at 180 minutes, and at follow-up (4-8 days after study day)
  Concentration of C-reactive protein in plasma
Experienced adverse effects post infusion | At 180 minutes.
  Number of experienced adverse effects as noted in a diary at end of each study day.
Experienced adverse effects during the four days following an infusion | During four days of follow-up after each study day.
  Number of experienced adverse effects as noted in a diary during four days of follow-up after each infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to GDPR regulations we are unable to share IPD with other researchers.